CLINICAL TRIAL: NCT01080079
Title: A Subject Blinded, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Iontophoretic Application of ETS Terbinafine Gel in Subjects With Distal Subungual Onychomycosis in the Great Toenail
Brief Title: Efficacy and Safety Study of Iontophoretic Application of Terbinafine Gel in Subjects With Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP-9
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Onychomycosis
Keywords: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A -Terbinafine HCl (Active Comparator): Terbinafine HCl
  Interventions: Drug: Terbinafine Hydrochloride
- Group B - Terbinafine HCl (Active Comparator): Terbinafine HCl
  Interventions: Drug: Terbinafine Hydrochloride
- Group C - Terbinafine HCl (Active Comparator): Terbinafine HCl
  Interventions: Drug: Terbinafine Hydrochloride
- Group D Terbinafine HCl (Active Comparator): Terbinafine HCl
  Interventions: Drug: Terbinafine Hydrochloride
- Group E (Active Comparator): Terbinafine HCl
  Interventions: Drug: Terbinafine Hydrochloride
- Group F - Placebo (Placebo Comparator): Placebo application
  Interventions: Other: Purified Water

INTERVENTIONS:
Drug: Terbinafine Hydrochloride — 4% w/w Terbinafine Hydrochloride Gel
  Arms: Group A -Terbinafine HCl; Group B - Terbinafine HCl; Group C - Terbinafine HCl; Group D Terbinafine HCl; Group E
Other: Purified Water — Purified Water
  Arms: Group F - Placebo

SUMMARY:
The purpose of this study is to determine if the iontophoretic application of terbinafine gel is safe and effective for teh treatment of distal subungual onychomycosis

ELIGIBILITY:
Inclusion Criteria:

- • Positive clinical findings for distal subungual onychomycosis as determined by clinical examination

* Must have a great toenail involvement with onychomycosis in ≥25-≤65% of the visible nail. (more than one nail maybe affected however only the index great toenail will be evaluated)
* Nail plate must be ≤ 3 mm thick.
* Must have a positive KOH and positive identification of a Dermatophyte via culture.
* Written informed consent must be obtained from the subject.
* Must be ≥ 18 and < 70 years of age, unless local laws dictate otherwise.
* Must agree to avoid any type of pedicure or application of any nail polish product or nail cosmetic to the toenails after the screening visit until the conclusion of the trial.
* Must agree to take measures to avoid pregnancy during the study period
* Must agree to avoid the use of oral or topical antifungals unless provided by the investigator for the relief of symptomatic (active clinical signs) tinea pedis which has occurred during the treatment / follow up phase of the study. (The treatment provided will be Lotrimin®).

Exclusion Criteria:

- • The presence of proximal subungual onychomycosis or white superficial onychomycosis

* Fungal involvement of the lunula or less than 2 mm of clear nail from the the proximal nail fold
* Subjects with psoriasis, eczema, symptomatic (with active clinical signs) interdigital or plantar tinea pedis, lichen planus, or other abnormalities (e.g. traumatized or dystrophic nails) that could result in a clinically abnormal nail or the investigator thinks the current condition will compromise the integrity of the trial
* Any presence of dermatophytoma or onychomycotic spikes
* Subjects with either uncontrolled diabetes mellitus or known diabetics on pharmaceutical therapy or those with no palpable pedal pulse
* Subjects with peripheral vascular disease
* Subjects who are immunosuppressed - those on chronic corticosteroid therapy (see below), with solid organ or bone marrow transplantation, cytotoxic chemotherapy within the previous 12 months (or planned within the next 12 months), or HIV infection.
* Use of topical antifungals e.g. (clotrimazole, ketoconazole, miconazole, oxiconazole (Oxistat®, Glaxo Smith Kline), sulconazole, naftifine (Naftin®, Merz), terconazole, econazole nitrate (Spectazole®, Ortho-McNeil), butoconazole ,Fluconazole, tolnaftate, haloprogin), Zeasorb-AF Ciclopirox (e.g. Penlac® Nail Lacquer, Sanofi-Aventis) and corticosteroids (e.g. hydrocortisone, betamethasone, fluticasone and mometasone) in the preceding 15 days of Day 1, on or immediately around the area under evaluation.
* Use of systemic corticosteroids within 30 days preceding Day 1
* Use of systemic antifungals in the preceding 120 days of Day 1 including - (terbinafine - (Lamisil®, Novartis), Itraconazole - (Sporanox®, Janssen), fluconazole- (Diflucan®, Pfizer), ketoconazole, miconazole, griseofulvin (Gris-PEG®, Pedinol), butoconazole, terconazole, potassium iodide,.
* Has used any investigational drug(s) within 30 days preceding Day 1, with the exception of investigational systemic antifungals (120 days))
* Is pregnant or is a nursing mother
* Is a woman of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Is < 18 years of age, unless local laws dictate otherwise.
* Suffers from a condition, which, in the opinion of the medical investigator, would compromise his/her safety and / or the quality of the data.
* Subjects with a pacemaker or automatic implantable cardioverter/defibrillator.
* Subjects with an implantable electronic device.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Clinical and Microbiological Improvement in nails vs placebo | 11 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - International Clinical Research, LLC, Sanford, Florida
  - Gwinnett Clinical Research Center, Inc, Snellville, Georgia
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Temple University Schoool of Podiatric Medicine, Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Endeavor Clinical Trials, PA, San Antonio, Texas
- Canada (2):
  - Mediprobe Research, Inc, London, Ontario
  - Lynderm Research, Inc, Markham, Ontario